CLINICAL TRIAL: NCT03971565
Title: Evaluation of the Redox Profiles of Healthy and Pathological B Cells in Patients With Chronic Lymphocytic Leukemia
Acronym: LLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-52; 2018-A02574-51 (Other: ID RCB)
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample of extra blood made as part of the care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic lymphocytic leukemia: Patient with a minimum period of 90 days without treatment
  Interventions: Biological: Blood sample 5 milliliter

INTERVENTIONS:
Biological: Blood sample 5 milliliter — The blood of the patients will be collected during their hospitalization of the hematology department participating in the research

SUMMARY:
In recent years, considerable progress has been made in understanding the biology of chronic lymphocytic leukemia (CLL), resulting in the emergence of new therapeutic agents that have significantly improved the long-term survival of patients. However, LLC is still considered an incurable disease.

Cytogenetic abnormalities are frequently found in this pathology. Some abnormalities are associated with a more aggressive disease and a poor prognosis. The deletion of chromosome 17p (del (17p)), in particular, makes leukemic cells more resistant to standard therapy. Chromosome 17p contains the Tumor Protein 53 gene (TP53) which encodes the tumor suppressor protein 53 (P53) protein. P53 plays a central role in the regulation of important cellular functions such as DNA damage response, cell cycle regulation, apoptosis, and drug sensitivity of chemotherapies. In patients with CLL, the loss of p53 function is a major factor of chemoresistance and is associated with an adverse prognosis. The deletion (17p) is observed in approximately 5 to 10% of patients with CLL. In contrast, mutations in the TP53 gene are observed in approximately 30% of patients with CLL. This means that about one-third of patients with CLL have p53 dysfunction. TP53 and / or del (17p) mutated LLC cells show marked mitochondrial dysfunction. This dysfunction is responsible for a deregulation of intracellular redox phenomena, leading to an increase in oxidative stress and an overproduction of reactive oxygen derivatives (ROS).

Dimethyl Ampal Thiolester (DIMATE) is an active, competitive and irreversible inhibitor of aldehyde dehydrogenases (ALDH) 1 and 3. In vitro, DIMATE eradicates human cells from acute myeloblastic leukemia (AML). In patients with CLL, current treatments, particularly effective, do not specifically target pathological B cells. This results in chronic B lymphopenia and hypogammaglobulinemias that provide severe long-term infections, which is the leading cause of death in patients with CLL.

Through this study, we will study, in vitro, the expression of ALDH 1, 3, 9 but also of glutathione (GSH) and ROS on tumor B lymphocytes and healthy patients carrying an LLC. Depending on the differences in expression observed, DIMATE could specifically eradicate leukemic lymphocyte cells by sparing healthy lymphocytes, a hypothesis that will be tested in vitro. A special evaluation will be made in patients with del (17) and / or TP53 mutation whose prognosis is still considered unfavorable despite new therapeutic advances.

ELIGIBILITY:
Inclusion Criteria:

* Major patient (greater than or equal to 18 years)
* Patients with 4 to 5 (or equivalent) grade 4 or 5 Matheol Score-confirmed chronic lymphocytic leukemia (CLL), whether prior to treatment or relapse
* For relapsed patients of their CLL, a minimum period of 90 days without treatment (including corticosteroids) compared to previous chemotherapy
* Patient having received the information and having given his non-opposition

Exclusion Criteria:

* Previous chemotherapy treatment outside of previous CLL therapy
* Active secondary cancer currently being treated with the exception of non-melanoma skin cancer or cervical cancer in situ
* Transformation into high grade lymphoma, Richter syndrome or pro-lymphocytic leukemia,
* Viral or fungal bacterial infection active at the time of screening Infection with human immunodeficiency virus,
* Medical or psychological condition that could interact with the ability to understand the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with chronic lymphocytic leukemia
Sampling Method: Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2019-03-19 (Actual); Primary Completion 2021-03-18 (Estimated); Study Completion 2021-03-18 (Estimated)

PRIMARY OUTCOMES:
Differentiate tumor B lymphocytes from normal B cells | 24 months
  Marker analysis is performed by flow cytometry to determine the expression of labeled aldehydes deshydrogenases (ALDH) molecules on tumor lymphocytes.
Differentiate tumor B lymphocytes from normal B cells | 24 months
  Marker analysis is performed by flow cytometry to determine the expression of labeled Gluthation (GSH) molecules on tumor lymphocytes.
Differentiate tumor B lymphocytes from normal B cells | 24 months
  Marker analysis is performed by flow cytometry to determine the expression of labeled reactive oxygen derivatives (ROS) molecules on tumor lymphocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assitance Publique Hôpitaux de Marseille
Locations (1):
- Assitance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No